CLINICAL TRIAL: NCT04077788
Title: Change of Range of Motion of TMJ After Correction of Pelvic a Symmetry in Women With Cyclic Pelvic Pain
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, rovan mohamed saad elbesh, Doctor, Misr University for Science and Technology
Other Study IDs: P.T.REC/012/001889
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group (group A):: It consisted of fifteen subjects who received muscle energy technique (Mitchell relaxation osteopathic technique). Two sessions per cycle for three cycles before menstruation by one week and after the end of menstruation by one week. In addition to their medical treatment non-steroidal anti-inflammatory drugs (NIAIDS).
  Interventions: Other: muscle energy technique
- control group (group B):: It consisted of fifteen subjects who took their medical treatment only (non-steroidal anti-inflammatory drugs (NIAIDS)).
  Interventions: Other: muscle energy technique

INTERVENTIONS:
Other: muscle energy technique — Muscle energy technique:
  1. Application of MET for bone of pelvis:
     I) Pubis:
     1. Cranial Os pubis.
     2. Caudal os pubis.
     II) ileum:
     1. Anterior ileum.
     2. Posterior ileum.
     3. External Rotation (In flare) Lesion.
     4. Internal Rotation (Out flare) Lesion.
     III) sacrum:
     1. Forward torsion of sacrum.
     2. Backward torsion of sacrum.
  2. Muscle energy technique for specific muscles of pelvis and spine:
     1. Stretch of the Psoas Major.
     2. Stretch of the paravertebral muscle.
     3. Stretch of the piriforms.

SUMMARY:
Clinical experiences have shown that significant pain regression during a menstrual cycle has been often achieved by the use of spinal manipulative therapy (SMT) indicated in women with primary dysmenorrhea with coexisting functional disorders of lumbosacral (LS) spine. Namely, by activation of the nociceptive and vegetative system, LS spine disorders, before all segmental dysfunction and degenerative changes, can induce referred pain and reflex disturbances of pelvic organs (somatovisceral reflexes). Since significant improvement or disappearance of pain during a menstrual cycle is often achieved with adequate therapy of coexisting vertebral disorders in women with primary dysmenorrhea, it is important to recognise latent or manifest vertebral disorders in dysmenorrheic women using clinical examination (Grgić, 2009).

ELIGIBILITY:
Inclusion criteria:

* The age of the participants will be ranged from 25 to 35 years.
* Their body mass index will be ranged from 20 to 25 kg/m2.
* They will have regular menstrual cycle.
* They will not receive any hormonal therapy or taking any regular drugs.

Exclusion criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Pelvic inflammatory diseases.
* Any pelvic pathological condition

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the participants will be divided randomly into two groups equal in numbers study group (group A) and control group (group B).
  • Study group (group A): It will consist of fifteen subjects who will receive osteopathic technique six treatment ( sessions) around three cycles two treatment every month first treatment after the end of menstruation.second treatment before the next cycle. In addition to their medical treatment if needed non-steroidal anti-inflammatory drugs (NIAIDS).
  • Control group (group B): It will consist of fifteen subjects who will reeive sham treatment,will take their medical treatment only non-steroidal anti- inflammatory drugs (NIAIDS) if needed.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Weight-Height Scale | 3 months
  It will be used for measuring the body weight and height of each patient participating in the study to calculate the patient's body mass index (BMI).
  Body mass index (BMI) = Weight (Kg
Visual analogue scale (VAS) | 3 months
  ain will be assessed by visual analogue scale. It is 10 cm horizontal line with one end described as (no pain=0) and other end (worst pain=10). It was considered a valid way for assessing pain. It allowed graphic representation and numerical analysis of collected data (Boonstra et al., 2008) (Appendix III).
Menstrual Distress Questionnaire (MDQ) | 3 months
  The MDQ is a 46-item self-report inventory for use in the assessment and treatment of premenstrual and menstrual symptoms. The MDQ can distinguish cyclical from noncyclical changes in physical symptoms, mood and behavior, and arousal.
jaw movement | 3 months
  Maximal vertical mouth opening (MIO):
  From sitting position, with the use of the calliper, the distance between the incisal edges along the midline of the upper and lower central incisors without pain was measured, by placing one end of the poley gauge against the incisal edge of one of the upper central incisors, and the other end against the incisal edge of the opposing lower incisor.
  The distance recorded in millimeters, the subjects was instructed to" open your mouth as wide as possible without causing pain or discomfort". The poley gauge was sterilized with antiseptic solution before and after each measur

CONTACTS AND LOCATIONS:
Locations (1):
- Rovan Elbesh, Giza, Egypt